CLINICAL TRIAL: NCT05156034
Title: A Randomized, Placebo-Controlled, Double-blind, Multiple Dose, Phase 1 Study to Evaluate the Safety, Tolerability, and Pharmacokinetics Following Intravenous Administration of SRK-001 in Healthy Participants
Brief Title: A Multiple Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of SRK-001 in Healthy Participants
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Due to occurrence of eye related adverse events.
Sponsor: Sarkana Pharma Inc (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SRKMD-2021; 2021-003991-15 (EudraCT Number)
Record Dates: First submitted 2021-11-16; First posted 2021-12-14 (Actual); Last update posted 2023-03-13 (Actual); Status verified 2023-03

CONDITIONS: Healthy Participants

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- SRK-001- Dose 1 (Experimental): Participants will receive intravenous (IV) SRK-001 every 2 weeks (Q2W) for 4 doses.
  Interventions: Drug: SRK-001
- SRK-001- Dose 2 (Experimental): Participants will receive IV SRK-001 every 4 weeks (Q4W) for 2 doses.
  Interventions: Drug: SRK-001
- SRK-001- Dose 3 (Experimental): Participants will receive IV SRK-001 Q2W for 4 doses.
  Interventions: Drug: SRK-001
- Placebo (Placebo Comparator): Participants will receive IV placebo Q2W for 4 doses or Q4W for 2 doses.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SRK-001 — Participants will receive IV doses of SRK-001.
  Arms: SRK-001- Dose 1; SRK-001- Dose 2; SRK-001- Dose 3
Drug: Placebo — Participants will receive IV doses of placebo.
  Arms: Placebo

SUMMARY:
The purpose of the study is to evaluate safety, tolerability, and pharmacokinetics (PK) of SRK-001 in Healthy Participants.

ELIGIBILITY:
Inclusion Criteria:

* Participants who have clinical chemistry laboratory values within the acceptable range for the population, as per the investigator judgment
* Body mass index of 18 to 32 kilogram (kg)/ square meter (m^2)
* Healthy male participants

  1. Nonvasectomized male participants must agree to abstain from sexual intercourse or use a condom as well as 1 additional highly effective method of contraception (less than [<]1 percent [%] failure rate) or effective method of contraception with all sexual partners of childbearing potential during the study and for 90 days following the last dose of study intervention
  2. Must agree not to donate sperm from start of dosing until 90 days beyond the last dose of study intervention
  3. No restrictions are required for a vasectomized male
* Healthy female participants of childbearing potential who have a fertile male sexual partner must be willing and able to practice effective contraception from screening to 90 days after the last dose of the study intervention. Sexually active participants must use a combination of 2 of the following methods of contraception, including at least 1 so-called 'barrier' method:

  1. hormonal contraceptives (oral, transdermal patches, vaginal, or injectable)
  2. intrauterine device with or without hormones
  3. condom, diaphragm, or cervical cap ('barrier' method)
  4. sexual abstinence, and
  5. vasectomized partner
* Has been fully vaccinated for COVID-19 with the last dose of vaccine administered at least 3 weeks prior to study intervention administration

Exclusion Criteria:

* For at least 30 days prior to randomization, participants must have no symptoms and/or signs of confirmed or suspected infection (including COVID-19) and must have completed any appropriate anti-infective treatment
* Have any concomitant systemic disorder, human immunodeficiency virus (HIV) infection, current infection with hepatitis B virus (HBV) (that is, positive for hepatitis B surface antigen and/or polymerase chain reaction positive for HBV DNA, hepatitis C virus (HCV) (that is, positive for HCV ribo nucleic acid[RNA]), symptomatic herpes zoster within 6 months prior to screening, an eye condition currently requiring treatment for trauma, contact allergy, postsurgical, or conjunctivitis that may interfere with eye evaluations, active or latent tuberculosis (TB)
* Are currently enrolled in or have participated in greater than (>) 4 clinical trials in the past 12 months involving a study intervention or off-label use of a drug or device, or any other type of medical research judged not to be scientifically or medically compatible with this study or have received a. any nonbiologic IP within 30 days or 5 half-lives (whichever is longer) of their baseline (Day -1) visit, or b. any biologic IP within 3 months or 5 half-lives (whichever is longer) of their baseline (Day -1) visit
* Have an average weekly alcohol intake that exceeds 21 units per week (males) or 14 units per week (females) or are unwilling to stop alcohol consumption from 48 hours prior to each dosing (1 unit = 12 ounce [oz] or 360 milliliter [mL] of beer; 5 oz or 150 mL of wine; 1.5 oz or 45 mL of distilled spirits)
* Drug abuse in the past 12 months and/or show positive findings on drug screening unless they were prescribed by a physician (for example, benzodiazepines)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2021-12-21 (Actual); Primary Completion 2022-09-05 (Actual); Study Completion 2022-09-05 (Actual)

PRIMARY OUTCOMES:
Number of Participants with One or More Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Event(s) (SAEs) | Baseline through final follow-up at approximately Day 155
  Number of participants with one or more TEAEs and SAEs will be reported in the adverse events module.

SECONDARY OUTCOMES:
Area Under the Concentration Versus Time Curve During a Dosing Interval (AUC0-tau) at Steady State | Day 1 (End of the infusion [EOI]) up to Day 155 post EOI
  Pharmacokinetics (PK) after single and multiple IV dosing.
Half-Life (t1/2) | Day 1 (EOI) up to Day 155 post EOI
  PK after single and multiple IV dosing.
Concentrations at End of Infusion (Cmax) | Day 1 (EOI) up to Day 155 post EOI
  PK after single and multiple IV dosing.
Concentrations at End of Dosing Interval (Ctrough) | Day 1 (EOI) up to Day 155 post EOI
  PK after single and multiple IV dosing.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Sarkana Pharma Inc
Locations (1):
- PRA Health Sciences, Groningen, Netherlands